CLINICAL TRIAL: NCT02325804
Title: Effect of Specific Diet and Circuit-based Exercise on Weight and/or Fat Loss
Brief Title: Effect of Specific Diet and Physical Activity on Weight and/or Fat Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slovak Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Adela Penesova, MD, PhD, Biomedical Center of Slovak Academy of Sciences, Institute of clinical and translational research, Slovak Academy of Sciences
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: FEXE- 11/2014
Record Dates: First submitted 2014-12-05; First posted 2014-12-25 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Obesity
Keywords: overweight and obesity; adipose tissue; weight loss program; low-calorie diet; circuit-based exercise; metabolic cardiovascular syndrome
MeSH Terms: conditions — Obesity; Overweight; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional lifestyle counseling (Active Comparator): Randomized, open label study to assess effect of 8 weeks of Conventional lifestyle counseling (low calorie diet and exercise) on body composition, physical fitness, and metabolic parameters
  Interventions: Behavioral: Lifestyle Counseling
- Unconventional lifestyle counseling (Active Comparator): Randomized, open label study to assess effect of 8 weeks of unconventional lifestyle counseling (low calorie "metabolic stairs" diet and circuit-based exercise) on body composition, physical fitness, and metabolic parameters
  Interventions: Behavioral: Lifestyle Counseling

INTERVENTIONS:
Behavioral: Lifestyle Counseling — In both arms life style counseling: Low calorie diet- 30% reduction of weight maintenance calories (TDEE); and recommended moderate exercise 3 times per week 45 minutes.

SUMMARY:
The main purpose of this study is to assess metabolic effects (decreased amount of body fat content, insulin sensitivity and lipid profile improvement) of weight loss intervention based on specific life style counseling (low calorie "metabolic stairs" diet and circuit-based exercise in a comparison to conventional diet and exercise. The main hypothesis is that more significant beneficial metabolic effects will have specific life style counseling effect than conventional diet and exercise. The main purpose of this study is to assess above mentioned metabolic changes before and after 6-8 weeks of weight loss intervention.

The investigators will also study the following:

1. The impact of life style counseling induced weight and/or fat loss on physical fitness
2. The impact of life style counseling induced weight and/or fat loss on metabolic parameters (e.g. insulin sensitivity, lipid profile, ect.)

DETAILED DESCRIPTION:
I

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* BMI≥25 kg/m2

Exclusion Criteria:

* Thyroid disease
* Chronic diseases(rheumatic,liver, kidney, pulmonary, etc. diseases) have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease, or diabetes;
* chronic infections
* show evidence of malignancy
* be women who are pregnant, nursing
* medical treatment except allergy medicines
* tobacco, alcohol or drug addiction

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
A Body weight change after specific weight loss intervention | 8 weeks
  To assess the body composition changes (fat-free mass and fat mass (in kg)).

SECONDARY OUTCOMES:
Metabolic parameters | 8 weeks
  * Insulin sensitivity
  * Total, HDL, LDL, small dense-LDL cholesterol levels

CONTACTS AND LOCATIONS:
Overall Officials: Adela Penesova, MD, PhD, Principal Investigator — Biomedical center, Slovak Academy of Sciences, Institute of clinical and translational researchBratislava, 833 06, SLOVAKIA
Locations (1):
- Biomedical Center, Slovak Academy of Sciences, Institute of clinical and translational reasearch, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Balaz M, Vician M, Janakova Z, Kurdiova T, Surova M, Imrich R, Majercikova Z, Penesova A, Vlcek M, Kiss A, Belan V, Klimes I, Olejnik J, Gasperikova D, Wolfrum C, Ukropcova B, Ukropec J. Subcutaneous adipose tissue zinc-alpha2-glycoprotein is associated with adipose tissue and whole-body insulin sensitivity. Obesity (Silver Spring). 2014 Aug;22(8):1821-9. doi: 10.1002/oby.20764. Epub 2014 Apr 22. PMID 24753506
- [Background] Penesova A, Radikova Z, Vlcek M, Kerlik J, Lukac J, Rovensky J, Imrich R. Chronic inflammation and low-dose glucocorticoid effects on glucose metabolism in premenopausal females with rheumatoid arthritis free of conventional metabolic risk factors. Physiol Res. 2013;62(1):75-83. doi: 10.33549/physiolres.932359. Epub 2012 Nov 22. PMID 23173679
- [Background] Penesova A, Venti CA, Bunt JC, Bonfiglio SM, Votruba SB, Krakoff J. Short-term isocaloric manipulation of carbohydrate intake: effect on subsequent ad libitum energy intake. Eur J Nutr. 2011 Sep;50(6):455-63. doi: 10.1007/s00394-010-0152-5. Epub 2010 Dec 17. PMID 21165629
- [Background] Penesova A, Cizmarova E, Belan V, Blazicek P, Imrich R, Vlcek M, Vigas M, Selko D, Koska J, Radikova Z. Insulin resistance in young, lean male subjects with essential hypertension. J Hum Hypertens. 2011 Jun;25(6):391-400. doi: 10.1038/jhh.2010.72. Epub 2010 Jul 15. PMID 20631738
- [Background] Penesova A, Bunt JC, Bogardus C, Krakoff J. Effect of paternal diabetes on pre-diabetic phenotypes in adult offspring. Diabetes Care. 2010 Aug;33(8):1823-8. doi: 10.2337/dc10-0664. Epub 2010 Jun 2. PMID 20519666
- [Background] Eckertova M, Krskova K, Penesova A, Radikova Z, Zlnay D, Rovensky J, Zorad S. Impaired insulin secretion and uptake in patients with diffuse idiopathic skeletal hyperostosis. Endocr Regul. 2009 Oct;43(4):149-55. PMID 19908933
- [Background] Penesova A, Radikova Z, Cizmarova E, Kvetnansky R, Blazicek P, Vlcek M, Koska J, Vigas M. The role of norepinephrine and insulin resistance in an early stage of hypertension. Ann N Y Acad Sci. 2008 Dec;1148:490-4. doi: 10.1196/annals.1410.036. PMID 19120146
- [Background] Ukropec J, Penesova A, Skopkova M, Pura M, Vlcek M, Radikova Z, Imrich R, Ukropcova B, Tajtakova M, Koska J, Zorad S, Belan V, Vanuga P, Payer J, Eckel J, Klimes I, Gasperikova D. Adipokine protein expression pattern in growth hormone deficiency predisposes to the increased fat cell size and the whole body metabolic derangements. J Clin Endocrinol Metab. 2008 Jun;93(6):2255-62. doi: 10.1210/jc.2007-2188. Epub 2008 Mar 11. PMID 18334583
- [Background] Skopkova M, Penesova A, Sell H, Radikova Z, Vlcek M, Imrich R, Koska J, Ukropec J, Eckel J, Klimes I, Gasperikova D. Protein array reveals differentially expressed proteins in subcutaneous adipose tissue in obesity. Obesity (Silver Spring). 2007 Oct;15(10):2396-406. doi: 10.1038/oby.2007.285. PMID 17925465
- [Background] Jurkovicova D, Sedlakova B, Riecansky I, Goncalvesova E, Penesova A, Kvetnansky R, Krizanova O. Cardiovascular diseases and molecular variants of the renin-angiotensin system components in Slovak population. Gen Physiol Biophys. 2007 Mar;26(1):27-32. PMID 17579251
- [Background] Penesova A, Cizmarova E, Kvetnansky R, Koska J, Sedlakova B, Krizanova O. Insertion/deletion polymorphism on ACE gene is associated with endothelial dysfunction in young patients with hypertension. Horm Metab Res. 2006 Sep;38(9):592-7. doi: 10.1055/s-2006-951307. PMID 16981142
- [Background] Penesova A, Rovensky J, Zlnay M, Dedik L, Radikova Z, Koska J, Vigas M, Imrich R. Attenuated insulin response and normal insulin sensitivity in lean patients with ankylosing spondylitis. Int J Clin Pharmacol Res. 2005;25(3):107-14. PMID 16366418
- [Background] Penesova A, Radikova Z. Comparison of insulin sensitivity indices calculated from standard 3-sampled and frequently sampled oral glucose tolerance test. Endocr Regul. 2004 Dec;38(4):167-71. PMID 15841797
- [Derived] Nechalova L, Bielik V, Hric I, Babicova M, Baranovicova E, Grendar M, Koska J, Penesova A. Gut microbiota and metabolic responses to a 12-week caloric restriction combined with strength and HIIT training in patients with obesity: a randomized trial. BMC Sports Sci Med Rehabil. 2024 Dec 5;16(1):239. doi: 10.1186/s13102-024-01029-7. PMID 39639405
- [Derived] Kubanova L, Bielik V, Hric I, Ugrayova S, Soltys K, Radikova Z, Baranovicova E, Grendar M, Kolisek M, Penesova A. Gut Microbiota and Serum Metabolites in Individuals with Class III Obesity Without Type 2 Diabetes Mellitus: Pilot Analysis. Metab Syndr Relat Disord. 2023 Jun;21(5):243-253. doi: 10.1089/met.2022.0071. Epub 2023 Apr 20. PMID 37083403
- [Derived] Bajer B, Radikova Z, Havranova A, Zitnanova I, Vlcek M, Imrich R, Sabaka P, Bendzala M, Penesova A. Effect of 8-weeks intensive lifestyle intervention on LDL and HDL subfractions. Obes Res Clin Pract. 2019 Nov-Dec;13(6):586-593. doi: 10.1016/j.orcp.2019.10.010. Epub 2019 Dec 2. PMID 31806470